CLINICAL TRIAL: NCT00844246
Title: Translating Evidence Based Developmental Screening Into Pediatric Primary Care ( Aims 2 and 3 )
Brief Title: Translating Evidence Based Developmental Screening Into Pediatric Primary Care
Acronym: TEDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2008-9-6124
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Developmental Delays
Keywords: Developmental delays; Early intervention services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SRS (Experimental): School Readiness Specialist (SRS) will administer the screening questionnaire to the subject during the intervention period, at the subject's 9, 18, 24 and 30 month visits. They will then see their PCP for a well child visit in which the results of the test will be interpreted, developmental counseling and/or anticipatory guidance provided as per usual care. EI (Early intervention) referral will be completed, at the discretion of the providers, if the subject fails the developmental screen or the caregivers raise a specific concern about the child's development.
  Interventions: Other: Developmental screening using ASQ and MCHAT
- Provider (Experimental): Primary Care Physician (PCP) will do the developmental screening at the subject's 9, 18, 24 and 30 month well child visits. Once the screening questionnaire is complete the PCP will then score the screening tool and interpret the test results. Developmental counseling and/or anticipatory guidance will be provided, as per usual care. EI (Early intervention) referral will be completed, at the discretion of the providers, if the subject fails the developmental screen or the caregivers raise a specific concern about the child's development.
  Interventions: Other: Developmental screening using ASQ and MCHAT
- Routine (No Intervention): Subjects randomized to routine surveillance will receive routine preventive care as well as developmental surveillance at all well child visits, including the 9, 18, 24 and 30 month visits. EI referral will be completed, at the discretion of the provider, if the PCP observes a developmental delay during surveillance or the caregivers raise a specific concern about the child's development.

INTERVENTIONS:
Other: Developmental screening using ASQ and MCHAT — In the SRS intervention arm subjects will complete developmental screening tools with a school readiness specialist at their 9, 18, 24 and 30 month well child visits and then complete their well child visit with their primary care clinician to discuss the results.
  Arms: SRS
Other: Developmental screening using ASQ and MCHAT — Subjects who are randomized to PCP arm will be screened for developmental delays by their Primary Care Clinician at their 9, 18, 24 and 30 month well child visits. The corresponding screening tools may be mailed to the study participants 2 weeks before the scheduled well child visits. Those who do not complete the screening tools or those who did not receive them in the mail will then complete the questionnaire in the office prior to seeing their doctor or with their doctor. The PCP will then score the screening tool and interpret the test results. Developmental counseling and/or anticipatory guidance will be provided, as per usual care. EI referral will be completed, at the discretion of the provider with the approval of the caregiver , if the subject fails the developmental screen or the caregivers raise a specific concern about the child's development.
  Arms: Provider

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability and effectiveness of implementing the American Academy of Pediatrics (AAP's) recommendation that clinicians provide developmental surveillance at all well child visits and institute developmental screening at critical developmental periods in childhood, namely at 9, 18, 24 and 30 months of age.

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility, acceptability and effectiveness of implementing the AAP's recommendation that clinicians provide developmental surveillance at all well child visits and institute developmental screening at critical developmental periods in childhood, namely at 9, 18, 24 and 30 months of age. The study will also examine its acceptance by pediatric practices, its adoption and adaptation in urban pediatric practices, and the effectiveness of a developmental screening protocol that conforms to the AAP and Maternal and Child Health Bureau (MCHB) recommendations compared with that of developmental surveillance alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age birth to 30 months of age by the start of the intervention phase.
2. Child's Primary Care Physician has consented to participate in the study
3. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Premature Infants (less than 36 weeks of gestation)
2. Children with prior identified developmental delay.
3. Children with major congenital anomalies/genetic disorders
4. Children placed in foster care

Max Age: 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2314 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for this study will be the percentage of children enrolled in the study who are identified as having a developmental delay. | We assessed this between June to October 2010

SECONDARY OUTCOMES:
Percentage of children in the study who are referred to Early Intervention Services | We assessed this in June 2010
Percentage of children in the study who enroll in Early Intervention Services | We will assess this between June to October 2010
Percent of parents enrolled in the study who report as satisfied with the intervention | We assessed this between March and September 2010
Percent of providers enrolled in the study who report as satisfied with the intervention. | We will assess this between March and September 2010

CONTACTS AND LOCATIONS:
Overall Officials: James P Guevara, MD MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - CHOP - Primary Care Market Street, Philadelphia, Pennsylvania
  - CHOP Primary Care-University City, Philadelphia, Pennsylvania
  - CHOP Primary Care Center- Cobbs Creek, Philadelphia, Pennsylvania
  - CHOP Primary Care - South Philadelphia, Philadelphia, Pennsylvania